CLINICAL TRIAL: NCT05250635
Title: Analysis of Breath Sound During Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-11-006BC
Record Dates: First submitted 2022-02-15; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Thoracic Surgery
Keywords: double lumen endobronchial tube; stethoscope; fiberscope; electronic stethoscope

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent thoracic surgery: Patients underwent thoracic surgery and general anesthesia with usage of DLET are included. Those patients with abnormal breath sound, pulmonary disease or history of cardiothoracic surgery are excluded.
  Interventions: Device: electronic stethoscope

INTERVENTIONS:
Device: electronic stethoscope — It includes main machine and auscultation patch, which can stick on patient's body to collect and amplify breath sound.

SUMMARY:
In modern thoracic surgery, double-lumen endobronchial tube (DLET) is the first choice for intubation. One lung ventilation can be perfectly performed by DLET, with the benefit of maintaining adequate gas exchange and establishing great surgical field. Traditionally, we use stethoscope and fiberscope for DLET site evaluation. However, there are some concerns over traditional methods. Stethoscope evaluation can be subjective from person to person; fiberscope, on the other hand, can cause additional bronchial injury as it is an invasive procedure. We hope to utilize patches, also known as electronic stethoscope, which provide non-invasive and visualized spectrum information, to assist anesthesiologists evaluate DLET insertion site more precisely in patients undergo thoracic surgery.

DETAILED DESCRIPTION:
This is an observational study. We use electronic stethoscope, which stick on patient's anterior chest, to record breath sound after intubation. The soundtrack will then be transformed to visualized waveform, enabling us to analyze and compare with actual result confirmed by fiberscope.

ELIGIBILITY:
Inclusion Criteria:

* patients undergo thoracic surgery and general anesthesia using DLET

Exclusion Criteria:

* patients have no will to participate
* vulnerable groups, including physically disabled and mental diseased patients
* patients with abnormal breath sound, pulmonary disease or history of cardiothoracic surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergo thoracic surgery and general anesthesia using DLET
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Accuracy of DLET intubation | Intraoperative (Start record the first breath sound after intubation when supine. After changing patient's position to lateral decubitus, the second breath sound is recorded. The electronic stethoscope is retrieved before the operation starts.)
  By using electronic stethoscope to record breath sound, we can analyze visualized waveform and spectrum to predict probable site and depth of DLET. Then we use fiberscope for actual result. By comparing records of electronic stethoscope and fiberscope, we hope to find correlation between these two methods of evaluating appropriate intubation of DLET.

SECONDARY OUTCOMES:
Correlation of breath sound and airway pressure | Intraoperative (Start record the first breath sound after intubation when supine. After changing patient's position to lateral decubitus, the second breath sound is recorded. The electronic stethoscope is retrieved before the operation starts.)
  During collection of breath sound, we also record airway pressure showed on ventilator at the same time. Theoretically, elevated airway pressure can be seen if airway obstruction or inappropriate intubation is happening. We hope to find correlation between airway pressure and breath sound collected by electronic stethoscope, for possible earlier detection, diagnosis and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Kun Ting, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No